CLINICAL TRIAL: NCT06540508
Title: Application of Integrated Proteomic and Serum Metabolomic Analysis in Assessing the Efficacy and Prognosis of TACE Combined With Targeted Immunotherapy in Unresectable Hepatocellular Carcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yue Han, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC3651
Record Dates: First submitted 2024-07-21; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Biospecimen Retention: Samples With DNA — 1. Peripheral Blood Samples (2 mL of serum):Blood needs to be centrifuged within 2 hours of collection (3000rpm for 15 minutes, then serum centrifuged again at 10000rpm for 15 minutes; aliquot 200 µL/tube and store at -80°C).
  2. Fecal Samples (2-3g):Procedure: Deposit feces into a clean container, avoiding contamination from urine or toilet surfaces; collect feces from the middle to end of bowel movement, preferably from the inner middle portion using a sterile spoon; place the fecal sample into an EP tube; immediately store them at -80°C.
  3. Urine Samples(10 mL):Procedure: Centrifuge 10 mL of urine (4°C, 10000rpm, for 5 minutes); transfer the supernatant to appropriately numbered EP tubes and freeze rapidly in liquid nitrogen, then store at -80°C.
  4. Liver Tumor Tissue Samples:Pre-cool and rinse tissues with saline to remove blood and debris; rapidly freeze tissue samples in liquid nitrogen, or store at -80°C if liquid nitrogen is not available.
  Storage of Remaining Samples: -80°C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group 1: Patients considered to have effective treatment after TACE combined with targeted immunotherapy, as assessed by mRECIST.
- Observation group 2: Patients considered to have ineffective treatment after TACE combined with targeted immunotherapy, as assessed by mRECIST.

SUMMARY:
Application of Integrated Proteomic and Serum Metabolomic Analysis in Efficacy and Prognosis Assessment: A multi-omics analysis based on gut microbiota to evaluate the predictive value of microbial-derived proteins and metabolites on treatment efficacy and patient outcomes, developing non-invasive tools for treatment monitoring and prognostic prediction.

DETAILED DESCRIPTION:
This study is a prospective, observational study based on real-world data. It prospectively and continuously collects data from patients with unresectable hepatocellular carcinoma who have received TACE combined with targeted and immunotherapy as part of their routine diagnostic and treatment procedures. Patients are grouped based on treatment efficacy, and integrated proteomic and serum metabolomic analyses are conducted on samples before and during treatment to obtain clinical evidence from the real world.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically or clinically diagnosed with hepatocellular carcinoma (HCC).
* Classified as BCLC stage B/C, not suitable for surgical resection or liver transplantation.
* Planned or already receiving TACE combined with tiragolumab and first-line targeted therapy for liver cancer.
* Not participating in other clinical studies.
* Able to obtain imaging evaluation data and other clinical records during treatment.

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed hepatocellular-cholangiocarcinoma histology.
* Tumors involving the main portal vein or inferior vena cava.
* Use of antibiotics within one month before treatment.
* History of other malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable hepatocellular carcinoma who have received TACE combined with targeted and immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Differences in Macroproteomics and Serum Metabolomics Expression between Effective and Ineffective Treatment Groups. | Starting from the completion of treatment and evaluation for all patients, up to 6 months
  Using two-dimensional liquid chromatography to separate proteins and perform data independent acquisition (DIA) for tissue and macro proteome analysis. Qualitative and quantitative analysis of DIA data was performed using data analysis software Spectronaut, and statistical algorithms were used to obtain differentially expressed proteins in HCC tissue and macro proteome between the effective and ineffective treatment groups. At the same time, non targeted metabolomics analysis methods were used to perform metabolomics analysis on serum samples from two groups of patients.
Model for predicting the efficacy and prognosis of advanced HCC treatment | Within six months after the completion of treatment and evaluation for all patients.
  Perform pathway and biological function enrichment analysis of differentially expressed proteins through IPA, analyze signal pathways and interaction networks of different bacterial strains through Unipept software, and perform pathway and functional analysis of differential metabolites through MetaboAnalyst to further screen important biomarkers. By using machine learning methods and combining ROC curves to construct efficacy prediction and prognosis judgment models, the optimal biomarker combination is obtained, and a prediction model is established.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No